CLINICAL TRIAL: NCT06332560
Title: Pain in Endometriosis And the Relation to Lifestyle: Effectiveness of a Dietary Intervention and Cognitive Behavioral Therapy in Endometriosis-associated Pain
Brief Title: Pain in Endometriosis And the Relation to Lifestyle
Acronym: PEARL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Belgian Volition SRL (Unknown); ASSOCIATION OF PEOPLE WITH ENDOMETRIOSIS I AM 1 IN 10 (Unknown); Wageningen University and Research (Other); Endometriosis UK (Unknown); University College Cork (Other); SVEUCILISTE U ZAGREBU MEDICINSKI FAKULTET (Unknown); UNIWERSYTET MEDYCZNY W LUBLINIE (Unknown); University of Edinburgh (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Université Catholique de Louvain (Other); University Bonn (Unknown); Biopsychology (Unknown); Horizon Europe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL86247.091.24
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-12

CONDITIONS: Endometriosis; Adenomyosis
Keywords: endometriosis; pain; quality of life; immunology; anti-inflammatory diet; cognitive behavioral therapy; adenomyosis; diet; microbiome
MeSH Terms: conditions — Endometriosis; Adenomyosis; Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Standard care (control group) (No Intervention)
- Standard care and an anti-inflammatory diet (DI group) (Experimental)
  Interventions: Behavioral: Anti-inflammatory diet (DI)
- Standard care, anti-inflammatory diet and cognitive behavioral therapy (DI + CBT group) (Experimental)
  Interventions: Behavioral: Anti-inflammatory diet (DI); Behavioral: Cognitive behavioral therapy (CBT)
- Standard care and cognitive behavioral therapy (CBT group) (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- Healthy controls (No Intervention): Healthy controls without endometriosis

INTERVENTIONS:
Behavioral: Anti-inflammatory diet (DI) — 12-week personalized dietary advice based on the Dutch Dietary Guidelines under the guidance of a dietician.
  Other Names: DI
  Arms: Standard care and an anti-inflammatory diet (DI group); Standard care, anti-inflammatory diet and cognitive behavioral therapy (DI + CBT group)
Behavioral: Cognitive behavioral therapy (CBT) — Seven individual sessions led by a psychotherapist. The content of the CBT will be psycho-education regarding pain mechanisms and DI.
  Other Names: CBT
  Arms: Standard care and cognitive behavioral therapy (CBT group); Standard care, anti-inflammatory diet and cognitive behavioral therapy (DI + CBT group)

SUMMARY:
The goal of this clinical trial is to investigate the effect of an anti-inflammatory diet and cognitive behavioral therapy (CBT) on pain symptoms, health related quality of life and the effect on inflammatory characteristics in serum and menstruum samples as well as the effect on the gut and vaginal microbiome in women with endometriosis. In addition, we want to investigate the differences in stress (measured by hair cortisol levels), inflammatory markers in peripheral blood, menstrual effluent, and the vaginal and intestinal microbiome between persons without and with endometriosis. Participants will be randomized between standard care (control group), standard care and an anti-inflammatory diet intervention, or standard care, an anti-inflammatory diet intervention and CBT or CBT alone. Participants will follow an anti-inflammatory diet based on the Dutch Dietary Guidelines or CBT or a combination of both interventions for 12 weeks. They will receive personalized dietary advice from a dietician and recipes will be available. cognitive behavioral therapy will be administered in a total of seven individual sessions led by a psychotherapist. The content of these sessions will be psycho-education regarding pain mechanisms (and diet).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of endometriosis via ultrasound, MRI or surgery*
* NRS pain score > 4*
* Age from 17 years
* Premenopausal status
* Body Mass Index (BMI) 18-30 kg/m2
* Ability to understand the explanation about the diet intervention (DI) and CBT*
* Willing to follow the DI*
* Willing to continue their use of food supplements
* Willing to undergo CBT*
* Willing to collect menstrual effluent, and therefore willing to have two stop weeks from hormonal contraception (if applicable) during the study period.

Exclusion Criteria:

* Recurrent miscarriages (> 2)
* Eating disorder
* Diagnosed with Crohn's disease, Ulcerative Colitis, short bowel syndrome or another chronic inflammatory disease
* Self-reported celiac disease
* Vegan diet
* Smoking
* Use of immunosuppressive or psychotropic medication
* Score on FFQ > 120
* Diagnosed with severe mental disorder currently requiring treatment by psychiatrist
* NRS average score below 4 during the last month
* Participation in another intervention study
* Unable to speak Dutch or to understand the intervention
* Need for surgery during the participation in the study
* Serious pain (NRS > 4) from other origin than endometriosis
* Pregnant
* Scalp hair shorter than 4 cm

  * Only applicable to patients with endometriosis

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — persons assigned female at birth
Enrollment: 250 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Pain intensity assessed by the Numerical Rating Scale | 3 months
  The Numerical Rating Scale (NRS) ranges from 0 (no pain) to 10 (unbearable pain), and is the most commonly used subjective measure to assess pain intensity. Patients will score there estimated average pain intensity and there highest pain intensity of the previous 7 days.
  Minimum value: 0 Maximum value: 10 Higher score indicates a higher level of pain intensity.

SECONDARY OUTCOMES:
Change in health related quality of life assessed by the Endometriosis Health Profile 30 | 3 months
  The Endometriosis Health Profile 30 (EHP-30) is a disease-specific QoL questionnaire which is validated for use in endometriosis patients and measures the impact of the disease on physical, mental and social aspects of life.
  The EHP-30 is not a numerical scale.
Change in general quality of llife assessed by the Short Form 36 | 3 months
  The Short Form 36 (SF-36) is a multipurpose, general health survey which is applied to measure QoL on nine different domains: physical functioning, social functioning, role limitations due to physical health, role limitations due to emotional problems, emotional well-being, vitality, pain, general health, and health change.
  The SF-36 is not a numerical scale.
Change in inflammatory characteristics in menstruum | 3 months
  High-dimensional flow cytometry will be done to analyse immune cells such as T cells, B cells, monocytes, and macrophages. Also Naturel Killer (NK) cells will be analysed. Also in the menstruum, markers for (cluster of differentiation 56) CD56, (cluster of differentiation antigen 16) CD16, (killer immunoglobulin receptors)) KIR and (natural cytotoxicity receptors) NCR, and activation markers such as CD69 will be characterised.
Change in inflammatory charecteristics in peripheral blood | 3 months
  High-dimensional flow cytometry will be done to analyse immune cells such as T cells, B cells, monocytes, and macrophages. Also NK cells will be analysed. Previous studies have described a key role for NK cells in endometriosis. A decreased percentage of NK cells was observed in peritoneal fluid of endometriosis patients compared to HC (Hoogstad-vanEvert et al., 2018 ). For in depth NK cell characterisation we will include markers for CD56, CD16, KIR (killer immunoglobulin receptors) and NCR (natural cytotoxicity receptors), and activation markers such as CD69.
Change in soluble factors in plasma | 3 months
  Analysed with the Olink Proteomics 96 inflammatory panel and Luminex multiplex assay for important soluble factors in endometriosis, i.e. IFNy, TNFα, TNFβ, IL1, IL2, IL6, IL8, IL12 and IL15, VEGF, Granzyme B, and perforin.
Change in the composition of vaginal and intestinal microbiome | 3 months
  Through 16S sRNA gene profiling the microbiome composition of faecal samples and vaginal swabs will be determined. Vaginal and faecal samples will be stored for later microbiome analysis if the the investigators see clear differences in inflammatory profiles after the dietary intervention.
Change in objective stress assessed by measuring scalp hair cortisol levels | 3 months
  Cortisol will be extracted from hair. The researcher will carefully collect a scalp hair sample of at least 0,5 cm thickness and sent these to the laboratory to analyze. The most proximal part represents the most recently grown piece of hair. Hair samples will be cut into a segment corresponding to the 4 cm closest to the scalp, reflecting cortisol secretion over the four months prior to sample collection. Cortisol extraction from hair will be carried out using an enzyme-linked immunoassay (ELISA).
Adherence and anti-inflammatory status of the diet | 3 months
  Diet quality will be assessed by the Eetscore. The Eetscore is a short (Food Frequency Questionnaire) FFQ, developed to assess the Dutch Healthy Diet 2015 (DHD2015) index. The questionnaire is composed of 40 questions assessing the frequency of consumption of food items. From the Eetscore FFQ, a DHD2015-index score can be calculated, indicating the diet quality of an individual.
  Ranges from 0 (unhealthy diet) - 160 (healthy diet).

OTHER OUTCOMES:
Change in sleep quality assessed by the PSQI | 3 months
  Sleep quality will be assessed by a self-rated questionnaire called (Pittsburgh sleep quality index) PSQI. This questionnaire contains 19 items, generating scores for seven different components. A general score can be obtained by adding up the scores of the seven components. Currently, PSQI is the most used tool in clinical and research practice assessing sleep quality.
  Minimum score: 0. Maximum score: 21. Higher scores indicate worse sleep quality.
Change in physical activity level assessed by the IPAQ-SF | 3 months
  Physical activity level will be assessed in this study to minimise confounding. Participants will fill in the (International Physical Activity Questionnaire Shor Form) IPAQ-SF, which is one of the most widely used self-report questionnaires assessing physical activity. This questionnaire assesses physical activity of the past seven days at four levels of intensity: vigorous, moderate, walking, and sitting.
  The IPAQ-SF sum score is expressed in PA Metabolic Equivalent of Task (MET)-minutes per day or week. A higher score corresponds to a physically more strenuous activity.
Change in subjective stress assessed by the PSS | 3 months
  Perceived stress will be measured using the Perceived Stress Scale (PSS), a 10-item validated psychological instrument for measuring nonspecific perceived stress. Items are designed to score how unpredictable, uncontrollable, and overloaded respondents find their lives.
  Minimum value: 10. Maximum value: 50. Higher score indicates a higher level of perceived stress.
Changes in pain cognitions assessed by the PASS | 3 months
  The Pain anxiety symptom scale (PASS) measures anxiety caused by pain. Questions are asked about feelings of fear of pain, cognitive anxiety, avoidance behaviour, and physiological anxiety symptoms.
  Minimum value: 0. Maximum value: 200. Higher score indicates a higher pain anxiety.
Changes in pain cognitions assessed by the PCS | 3 months
  The pain catastrophizing Scale (PCS) measures the degree of pain catastrophizing of the participant by measuring elements of helplessness and pessimism in relation to the ability to cope with the pain experience.
  Minimum value: 0. Maximum value: 52. Higher score indicates a higher level of catastrophizing
Changes in fatigue assessed by the CIS | 3 months
  The checklist Individual Strength (CIS) is a 20-item questionnaire addressing fatigue, concentration, motivation and activity over the past two weeks.
  The CIS is not a numerical scale.
Anti-inflammatory diet rating | At the end of the intervention (3 months), when completed the diet intervention
  At the end of the intervention period, participants will evaluate the anti-inflammatory diet with a rating on scale, and several general questions concerning the taste, cost, and feasibility.
  Minimum value: 1 Maximum value: 10. Higher scores indicates greater satisfaction with the diet.
Epigenetics | 3 months
  The global level of nucleosomes and the levels of nucleosome containing specific histone post-transcriptional modifications will be analyzed in menstrual effluent and/or K2-EDTA plasma samples from healthy patients (n=50) and from patients in the SC + DI and SC + DI + CBT group. DNA extraction from K2-EDTA plasma samples or from menstrual effluent, and DNA amount quantification and fragments length qualification Analysis of the samples will be performed using Nu.Q® immunoassays according to the instructions of the SME company Volition (Belgium), allowing for the quantification of specific nucleosome structures.
Untargeted general plasma metabolomics | 3 months
  To measure metabolites, to understand the impact of both interventions on metabolic pathways
Differences in inflammatory characteristics in menstruum and peripheral blood between patients with endometriosis and healthy controls | Baseline
  High-dimensional flow cytometry will be done to analyse immune cells such as T cells, B cells, monocytes, and macrophages. Also NK cells will be analysed. Previous studies have described a key role for NK cells in endometriosis. A decreased percentage of NK cells was observed in peritoneal fluid of endometriosis patients compared to HC (Hoogstad-vanEvert et al., 2018 ). For in depth NK cell characterisation we will include markers for CD56, CD16, KIR (killer immunoglobulin receptors) and NCR (natural cytotoxicity receptors), and activation markers such as CD69.
Differences in the composition of vaginal and intestinal microbiome in patients with endometriosis and healthy controls | Baseline
  Through 16S sRNA gene profiling the microbiome composition of faecal samples and vaginal swabs will be determined.
Differences in stress (measured by hair cortisol level) in patients with endometriosis and healthy controls | Baseline
  Cortisol will be extracted from hair. The researcher will carefully collect a scalp hair sample of at least 0,5 cm thickness and sent these to the laboratory to analyse. The most proximal part represents the most recently grown piece of hair. Hair samples will be cut into a segment corresponding to the 4 cm closest to the scalp, reflecting cortisol secretion over the four months prior to sample collection. Cortisol extraction from hair will be carried out using an enzyme-linked immunoassay (ELISA) (DRG Instruments GmbH, Marburg, Germany). Analysis of the samples will be performed according to the instructions of the ELISA kit manual at Biopsychology - TU Dresden (Germany).

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Jeroen Bosch Hospital (JBZ), 's-Hertogenbosch
  - Rijnstate Hospital, Arnhem
  - Amphia, Breda
  - Catharina Hospital, Eindhoven
  - Radboud University Medical Center, Nijmegen

IPD SHARING:
Plan to Share IPD: No